CLINICAL TRIAL: NCT06350708
Title: Can Remote Training of Paediatric Emergency Tracheostomy Simulation be Performed Using VR Technology?
Brief Title: Virtual Reality (VR) Paediatric Tracheostomy Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jonathan Abass, Principal Investigator, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-18304-33663; 336664 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Educational Study
Keywords: virtual reality; tracheostomy; training; paediatric

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Virtual reality (VR) tracheostomy educational tool — This is an unsupervised VR training packaged designed to train healthcare professionals and their students the management of the paediatric tracheostomy emergency.

SUMMARY:
This study aims to evaluate the use of an unsupervised virtual reality training tool. This tool is used to teach nurses, doctors and other healthcare workers and their students how to manage tracheostomy emergencies in children.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare student
* Clinical experience needed
* Healthcare staff
* Based at Manchester University Foundation Trust, or The University of Manchester

Exclusion Criteria:

* Not a healthcare student
* Not a healthcare student - have no clinical experience
* Not healthcare staff but working in the National Health Service
* Not based at Manchester University Foundation Trust, or The University of Manchester

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Performance in simulation (time to key specific intervention, time to completion of scenario, and number of correct interventions completed) | Measured at the beginning of study and 1 week.
  Test the improvement in simulated performance in a pre- and post-test method.
  Time to key specific intervention and total scenario times will be measured in seconds, with a smaller number indicating better performance.
  Number of correct interventions will be simple numerical with higher number indicating better performance.

SECONDARY OUTCOMES:
Knowledge using a bespoke knowledge multiple choice questionnaire adapted from a validated question bank. | Measured at the beginning of study,1 week and 4 weeks post intervention.
  Measurement of knowledge in a pre- and post-test method. The a higher score will indicate more knowledge. Minimum values are 0, maximum value of 23.
Participant satisfaction measured using a bespoke data collection tool. | 1 week post initiation of intervention
  Likert questionnaire
Virtual Reality Sickness | 1 week post initiation of intervention
  Measure of participant comfort using the validated Virtual Reality Sickness Questionnaire.
  Lower score is better. The score can range from 0-27.
Usability using the validated system usability scale | 1 week post initiation of intervention
  Measure of usability using the validated System Usability Scale
  Calculation of the score is complex, and will follow the guidance in the below academic work:
  https://www.researchgate.net/publication/228593520_SUS_A_quick_and_dirty_usability_scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbas JR, Younis N, Johnstone E, Rajai A, Isba R, Payton A, McGrath BA, Tolley N, Bruce IA. Use of virtual reality to remotely train healthcare professionals in paediatric emergency tracheostomy skills: protocol for a multi-centre, non-inferiority educational interventional study with historical controls. BMC Surg. 2025 Jan 15;25(1):25. doi: 10.1186/s12893-024-02736-1. PMID 39810190